CLINICAL TRIAL: NCT00821366
Title: Effective Aids Treatment and Support in the Free State (FEATS): Adherence and Nutritional Support for Effective and Sustainable Antiretroviral Treatment in Resource Constrained Settings
Brief Title: Effective Aids Treatment and Support in the Free State (FEATS)
Acronym: FEATS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre for Health Systems Research & Development, University of the Free State (Other)
Collaborators: World Bank (Other); Bank-Netherlands Partnership Programme (BNPP) (Unknown)
Responsible Party: Professor Frikkie Booysen, University of the Free State
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FEATS
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-01

CONDITIONS: HIV/AIDS; Food Insecurity; HIV Infections
Keywords: HIV/AIDS; Food security; treatment experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Nutritional Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Households including ARV patients who receive the ARV treatment and associated support provided as part of government's ARV treatment programme - ARV treatment only group
  Interventions: Drug: ARV treatment
- 2 (Active Comparator): Households including ARV patients who receive the ARV treatment and associated support provided as part of government's ARV treatment programme - ARV treatment and ARV peer adherence support group
  Interventions: Behavioral: ARV peer adherence support (PAS); Drug: ARV treatment
- 3 (Active Comparator): Households including ARV patients who receive the ARV treatment and associated support provided as part of government's ARV treatment programme - ARV treatment, ARV peer adherence support and nutritional support group
  Interventions: Behavioral: ARV peer adherence support (PAS); Dietary Supplement: Nutritional support; Drug: ARV treatment
- 4 (No Intervention): Randomly selected households from the general community served by the selected health facility, excluding households where someone is known to receive ARV treatment - comparison/control group

INTERVENTIONS:
Behavioral: ARV peer adherence support (PAS) — Adherence support provided during twice weekly visits to the patient by an experienced ART patients who received basic training in ARV peer adherence support
  Arms: 2; 3
Dietary Supplement: Nutritional support — Weekly delivery by peer adherence supporter (PAS) of two 400g cans of meatballs and spaghetti in tomato sauce
  Arms: 3
Drug: ARV treatment — Households including ARV patients who receive the ARV treatment and associated support provided as part of government's ARV treatment programme
  Arms: 1; 2; 3

SUMMARY:
The aim of this study is to investigate the benefits of ARV treatment to patients, to the family members of patients on ARV treatment, and to communities at large. The study also aims to investigate the impact of a peer adherence support and a nutritional intervention on measures of treatment success. To this end, 648 patients who had commenced ARV treatment in the past month at twelve selected health care facilities will be recruited into the study. In addition, 204 randomly sampled households from the communities served by the twelve selected clinics will be recruited into the study. Trained enumerators will at baseline conduct semi-structured interviews with patients and households. Following the baseline survey, patients recruited into the study will be randomly assigned to one of three groups:

* Patients receiving ARV treatment and the associated support currently provided in the public sector ARV treatment programme.
* Patients receiving (a) plus bi-weekly visits by an experienced ARV patient who has been trained as a peer adherence supporter
* Patients receiving (a) and (b) plus a weekly nutritional supplement in the form of two 400g cans of meatballs and spaghetti in tomato sauce The group of 'comparison' households comprises the fourth group. Trained enumerators will conduct follow-up interviews with all patients and households at approximately six- and at twelve-months respectively. In addition, the ARV coordinator and other providers working in the ARV treatment programme at each of the twelve selected health care facilities will be interviewed by trained enumerators, at baseline and again at six- and at twelve-months. Clinical data will be obtained from patient files at baseline and at completion of the study. Using these data, various outcomes of importance to the study will be compared between the four study groups, using experimental and non-experimental methods.

DETAILED DESCRIPTION:
The study has three main objectives, each with a set of more specific aims:

Objective 1: Present a broader view of treatment success

In order to achieve this objective, the study aims to:

* Investigate how access to antiretroviral treatment and to nutritional supplementation impacts labour productivity and time allocation of patients and other household members
* Investigate how access to antiretroviral treatment and to nutritional supplementation impacts household welfare
* Investigate how access to antiretroviral treatment and to nutritional supplementation impacts educational and health outcomes for children in households with patients on antiretroviral treatment

Objective 2: Develop a model of the determinants of treatment success

In order to achieve this objective, the study aims to:

* Determine how various individual, household and facility-level characteristics impact adherence to antiretroviral treatment, including access to a disability grant
* Determine how access to a peer adherence supporter and nutritional supplementation impacts adherence to antiretroviral treatment
* Estimate the cost-effectiveness of these interventions in enhancement in adherence, from both a fiscal and a social perspective

Objective 3: Understand the links between treatment and prevention

In order to achieve this objective, the study aims to:

* Determine how access to antiretroviral treatment impacts on the uptake of voluntary counselling and testing among members of households including patients on ARV treatment and among members of households in the general community
* Determine how access to antiretroviral treatment, to a peer adherence supporter and to nutritional supplementation impacts on the sexual behaviour of patients on antiretroviral treatment, their household members, and members of households in the general community

The study aims to investigate effective AIDS treatment and support in settings where free ARV treatment has been introduced already, with issues of scale-up and sustainability as a result representing an important issue. The study therefore is being conducted in twelve phase I ARV assessment sites in the Free State province, i.e. sites where ARV treatment first became available when the ARV treatment programme was launched in the Free State province in 2004/05.

1. Type of study The study is a prospective, cohort study with a patient, household, facility and provider survey component. The study has a social scientific focus, with a clinical component, and comprises two behavioural interventions.
2. Description of experimental design The study is a combination of a group time-series quasi-experimental design and a a variation of a double randomised consent design. The study comprises four groups of households, three of which include patients on ARV treatment (Figure 1). The provision of ARV treatment represents a quasi- or field experiment, while the peer adherence support and nutritional interventions represent a randomised-control experiment executed in accordance with a Zelen-type double randomised consent design. This study design is deemed appropriate given the fact that: blinding is not practicable or possible; the use of classical randomisation and informed consent procedures significantly threatens internal validity; the interventions are highly attractive; the control group receives standard care; the study focuses on a clinically relevant objective(s) and offers important new insights (Kaptchuk, 2001; MacLehose et al, 2001; Rains & Penzien, 2005).

   Figure 1: Experimental study design

   Group A: Households including ARV patients who receive the ARV treatment and associated support provided as part of government's ARV treatment programme Sample size: n~216]

   Group B: Households including ARV patients who receive the ARV treatment and associated support provided as part of government's ARV treatment programme PLUS Adherence support provided by a trained peer adherence supporter during twice weekly visits to the patient [Sample size: n~216]

   Group C: Households including ARV patients who receive the ARV treatment and associated support provided as part of government's ARV treatment programme PLUS Adherence support provided by a trained peer adherence supporter during twice weekly visits to the patient PLUS Nutritional supplementation: weekly delivery of two 400g cans of meatballs and spaghetti in tomato sauce by peer adherence supporter [Sample size: n~216]

   Group D: Randomly selected households from the general community served by the selected health facility, excluding households where someone is known to receive ARV treatment [Sample size: n~180]

   Sample size estimation:

   The sample size calculation for the arms of the study is based on the method proposed by Freedman (1982). The sample size estimation is based on the following assumptions:
   * The proportion of people showing an improvement in a specific outcome, are compared across two arms of the study at a time.
   * Attrition in the control group of comparison households is assumed to be minimal or none (since there is no ARV patient in the household), while attrition in the intervention arms (where ARV treatment is considered an intervention) is assumed to be much higher, given a reported mortality of 10% among ARV patients in the first months of treatment (Free State Department of Health, 2006).
   * The required sample sizes for a 4-equal-arms-at-end-of-study design were calculated taking into account the attrition rate of 17% in the three intervention groups and a ratio of 1 for the treatment: control arms at the end of the study is expected.
   * Assuming a two-tailed test with Type I error of 5%, Type II error of 10%, and at least 17% improvement in any outcome.

   The affordable sample size was 801 households with 177 for the control arm and 208 for each of the intervention arms. This sample is expected to yield statistically significant results for the analysis of all measures contemplated. Although the statistical power of the study design with this sample size can be considered good the sample size was rounded up to ~828 households, with ~180 households in the control arm and ~216 households in each of the intervention arms. This was done to represent multiples of 12 since the study will be conducted in 12 facilities.
3. Method of randomisation From among the ~648 ARV patients recruited into the study [~54/study site], individual patients will be assigned randomly to the control group [Group A; n~216] and to the two experimental arms of the study [Group B & C; n~216 each], using the relevant random sampling selection commands in version 10 of the Stata software programme.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* Eligible for public sector ARV treatment (CD4<200 and/or WHO stage 4)
* Commenced ARV treatment in past 4 weeks
* Patient resident in town/village where ART clinic located

Exclusion Criteria:

* HIV-negative
* Not eligible for public sector ARV treatment
* Had not commenced ARV treatment
* Commenced ARV treatment longer than one month ago
* Patient not resident in town/village where ART clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2007-10; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
CD4 count | 6-monthly
RNA viral load | 6-monthly
Haemoglobin | 6-monthly
self-reported adherence (CASE index) | 6-monthly
health-related quality of life (EQ-5D/EQ-VAS) | 6-monthly
anthropometrics | monthly to 6-monthly
food security (USDA scales) | 6-monthly
time allocation/physical activity levels | 6-monthly
household welfare | 6-monthly

SECONDARY OUTCOMES:
mental health (HADS/MHI scales) | 6-monthly
labour force participation | 6-monthly
employment status | 6-monthly
self-reported sexual behaviour | 6-monthly
school attendance/performance | 6-monthly

CONTACTS AND LOCATIONS:
Overall Officials: Frikkie LR Booysen, PhD, Study Director — University of the Free State
Locations (12):
- South Africa (12):
  - Batho clinic, Bloemfontein, Free State
  - MUCPP clinic, Bloemfontein, Free State
  - Tswelepele clinic, Bloemfontein, Free State
  - Refengkhotso clinic, Deneysville, Free State
  - Tshiame clinic, Harrismith, Free State
  - Itumeleng clinic, Jagersfontein, Free State
  - Phomolong clinic, Phomolong, Free State
  - Namahali clinic, Phuthaditjaba, Free State
  - Tseki clinic, Phuthaditjaba, Free State
  - Zamdela clinic, Sasolburg, Free State
  - Matjhabeng clinic, Welkom, Free State
  - Welkom clinic, Welkom, Free State

REFERENCES:
- [Derived] Bhargava A, Booysen FLR, Walsh CM. Health status, food insecurity, and time allocation patterns of patients with AIDS receiving antiretroviral treatment in South Africa. AIDS Care. 2018 Mar;30(3):361-368. doi: 10.1080/09540121.2017.1371665. Epub 2017 Sep 1. PMID 28862017